CLINICAL TRIAL: NCT01598415
Title: A Two Part Protocol to Assess, Using Double Blind Placebo Control, the Safety, Tolerability, and Pharmacokinetics of Ascending Single Doses of a New Intra-articular Administration Formulation of SAR113945 (IKK Inhibitor) Followed by Assessment of Efficacy, Safety, Tolerability and Pharmacokinetics of a Single Dose in Patients With Knee Osteoarthritis.
Brief Title: Safety of Single Doses of SAR113945 and Efficacy and Safety of a New Formulation Given Into the Knee in Osteoarthritis Patients / Part II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT12505; 2011-003232-31 (EudraCT Number); U1111-1124-5323 (Other: UTN); TDU11685/ACT12505 (Other: sanofi-aventis other study code)
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAR113945 (Experimental): TDU11685 selected dose
  Interventions: Drug: SAR113945
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAR113945 — Pharmaceutical form:Injection
  Route of administration: Intra-articular
  Arms: SAR113945
Drug: placebo — Pharmaceutical form:Injection
  Route of administration: Intra-articular
  Arms: Placebo

SUMMARY:
Study objectives:

* Part 1 TDU11685 To assess in patients with knee Osteoarthritis (OA), the safety, tolerability and pharmacokinetics (PK) of single intra-articular doses of SAR113945.
* Part 2 ACT12505 To assess in patients with knee OA, the efficacy, safety and tolerability of a single intra-articular dose of SAR113945.

DETAILED DESCRIPTION:
- Screening will be performed within 28 days of dosing. Following the single dose of study medication, the study period for each patient will be 168 days.

ELIGIBILITY:
Inclusion criteria :

Diagnosis of primary knee osteoarthritis, based upon the following:

* X-ray or Magnetic Resonance Imaging (MRI) evidence within the last 6 months for joint space narrowing and osteophyte formation
* Patients will be Kellgren and Lawrence classification II/III, and total Western Ontario McMaster (WOMAC) score 24 -72.
* Patients fulfilling the American College of Rheumatology Clinical and Radiographic criteria for Osteoarthritis.

Exclusion criteria:

* Patients younger than 40 years
* Women of child bearing potential.
* Women either sterilized for more than 3 months, or post-menopausal for more than 12 months. Menopause is defined as over age of 60 years or being amenorrheic for at least 2 years with plasma FSH level >30 IU/L.
* Secondary osteoarthritis: e.g., autoimmune disease, joint dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler's syndrome, joint infection, haemophilia, haemochromatosis, calcium pyrophosphate deposition disease, or neuropathic arthropathy.
* Presence of local skin abnormality at the affected knee joint.
* Intra-articular injection within 3 months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Womac Pain Score (5 items) | at 8 weeks

SECONDARY OUTCOMES:
Womac Pain Score (5 items) | during 24 weeks
Womac Total Score (24 items) | during 24 weeks
Womac Stiffness (2 items) | during 24 weeks
Womac Physical Function (17 items) | during 24 weeks
synovial fluid levels | during 24 weeks
Number of patients reporting Adverse Events of special interest: tolerability at the site of injection and in the knee + other events reported by the patient | during 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Germany (2):
  - Investigational Site Number 276001, Berlin
  - Investigational Site Number 276002, München